CLINICAL TRIAL: NCT04757194
Title: Machine Learning Assisted Differentiation of Low Acuity Patients at Dispatch: A Randomized Controlled Trial
Brief Title: Machine Learning Assisted Differentiation of Low Acuity Patients at Dispatch
Acronym: MADLAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Region Västmanland (Other)
Responsible Party: Principal Investigator, Hans Blomberg, Medical Director, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SVLC001
Record Dates: First submitted 2021-02-03; First posted 2021-02-17 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Groups of patients experiencing a resource constrained situation randomized 1:1 at time of inclusion to control/intervention arms
Who Masked: Investigator
Masking Description: Analyst masked to treatment group allocation in final analysis. Outcomes extracted algorithmically from databases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Calculation of risk assessment score by machine learning algorithm and display of risk assessment information to dispatch nurses. Staff encouraged but not required to comply with suggested ranking.
  Interventions: Diagnostic Test: openTriage - Alitis algorithm
- Control (No Intervention): Ambulance dispatch per standard of care

INTERVENTIONS:
Diagnostic Test: openTriage - Alitis algorithm — A machine learning algorithm (Gradient boosting) applied to structured data collected in the Alitis Clinical Decision Support system, patient demographics, and free-text notes.
  Arms: Intervention

SUMMARY:
BACKGROUND:

At Emergency Medical Dispatch (EMD) centers, Resource Constrained Situations (RCS) where there are more callers requiring an ambulance than there are available ambulances are common. At the EMD centers in Uppsala and Västmanland, patients experiencing these situations are typically assigned a low-priority response, are often elderly, and have non-specific symptoms. Machine learning techniques offer a promising but largely untested approach to assessing risks among these patients.

OBJECTIVES:

To establish whether the provision of machine learning-based risk scores improves the ability of dispatchers to identify patients at high risk for deterioration in RCS.

DESIGN:

Multi-centre, parallel-grouped, randomized, analyst-blinded trial.

POPULATION:

Adult patients contacting the national emergency line (112), assessed by a dispatch nurse in Uppsala or Västmanland as requiring a low-priority ambulance response, and experiencing an RCS.

OUTCOMES:

Primary:

1. Proportion of RCS where the first available ambulance was dispatched to the patient with the highest National Early Warning Score (NEWS) score

Secondary:

* Difference in composite risk score consisting of ambulance interventions, emergent transport, hospital admission, intensive care, and mortality between patients receiving immediate vs. delayed ambulance response during RCS.
* Difference in NEWS between patients receiving immediate vs. delayed ambulance response during RCS.

INTERVENTION:

A machine learning model will estimate the risk associated with each patient involved in the RCS, and propose a patient to receive the available ambulance. In the intervention arm only, the assessment will be displayed in a user interface integrated into the dispatching system.

TRIAL SIZE:

1500 RCS each consisting of multiple patients randomized 1:1 to control and intervention arms

ELIGIBILITY:
Inclusion Criteria:

* Identification of a resource constrained situation by ambulance director (i.e., 2 or more patients awaiting an ambulance response)
* Assigned priority 2A or 2B (Low-priority ambulance response) by dispatch nurse call-taker
* Valid Swedish personal identification number collected at dispatch
* Age >= 18 years

Exclusion Criteria:

* Relevant calls received more than 30 minutes apart
* Logistical factors (eg. the patients' geographical locations) affect the ambulance assignment decision
* On scene risk factors (eg. a patient is outdoors and risks hypothermia) or risk mitigators (eg. healthcare staff already on-scene with a patient) affect the ambulance assignment decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2499 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of RCS where the first available ambulance was dispatched to the patient with the highest National Early Warning Score (NEWS). | Upon ambulance response (Within 8 hours of dispatch)
  NEWS is a widely used and well-validated scoring algorithm based on objective patient vital signs, which are not causally dependent on the outcomes used to train the machine learning models investigated in this study. NEWS values will be based on the first set of vital signs obtained by ambulance nurses upon making contact with the patient. NEWS is measured on a 0-21 scale, with higher values corresponding to patients at higher risk for deterioration.

SECONDARY OUTCOMES:
Difference in composite outcome measure score between patients with immediate vs. delayed response. | Up to 30 days
  This measure investigates a composite score consisting of the outcomes used to train the machine learning models. The composite score is generated by identifying the following patient outcomes and assigning the corresponding weights:
  Abnormal intitial Arway/Breathing/Circulation findings by ambulance crew (4) Emergent (lights and sirens) transport to the hospital (2) Provision of prehospital interventions (1) Admission to in-patient care or mortality within 30 days (1)
  This results in a score from 0-8, with higher scores representing more
Difference in National Early Warning Score (NEWS) between patients with immediate vs. delayed response. | Upon ambulance response (Within 8 hours of dispatch)
  Per primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Hans Blomberg, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (2):
- Sweden (2):
  - Västmanland hospital Västerås, Västerås, Västmanland County
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Individual level data available upon reasonable request to authors after publication
Supporting Information: Study Protocol, Analytic Code
Time Frame: Upon publication
Access Criteria: Researchers with ethics board approved research plan

REFERENCES:
- [Background] Spangler D, Hermansson T, Smekal D, Blomberg H. A validation of machine learning-based risk scores in the prehospital setting. PLoS One. 2019 Dec 13;14(12):e0226518. doi: 10.1371/journal.pone.0226518. eCollection 2019. PMID 31834920
- [Background] Spangler D, Edmark L, Winblad U, Collden-Benneck J, Borg H, Blomberg H. Using trigger tools to identify triage errors by ambulance dispatch nurses in Sweden: an observational study. BMJ Open. 2020 Mar 19;10(3):e035004. doi: 10.1136/bmjopen-2019-035004. PMID 32198303
- See also: Source code for risk assessment tool used in intervention — https://github.com/dnspangler/openTriage

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT04757194/Prot_SAP_000.pdf